CLINICAL TRIAL: NCT06642636
Title: Intensive Care Unit-specific Virtual Reality As Preparation for ICU Admission in Lung Transplant Patients
Brief Title: ICU-VR Prior to ICU Admission
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Denzel Drop (Other)
Responsible Party: Sponsor-Investigator, Denzel Drop, MD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL87675.078.24
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Post Intensive Care Syndrome (PICS); PTSD - Post Traumatic Stress Disorder
Keywords: virtual reality; extended reality; intensive care; intensive care unit; intensive care units; critical care; lung transplantation; ICU-VR
MeSH Terms: conditions — postintensive care syndrome; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICU-VR (Experimental): Regarding the participants in the intervention group, an appointment will be scheduled with a nurse specialist of the department of pulmonology and a researcher to watch the ICU-VR intervention. During this appointment, patients will be allowed to watch the VR video as many times as desired.
  Interventions: Device: Intensive Care Unit-specific Virtual Reality
- Control (No Intervention): The control group will receive the usual care and no intervention.

INTERVENTIONS:
Device: Intensive Care Unit-specific Virtual Reality — The Intensive Care specific Virtual Reality (ICU-VR) film is designed so that patients received relevant and truthful information regarding their ICU treatment with the aim to reduce stress and anxiety. The final film lasts approximately 12 minutes. Real ICU nurses and ICU physicians re-enacting a typical day/treatment for a mock patient undergoing ICU treatment. The module will be watched via HMD-VR glasses (PICO G2 VR; Pico Technology, Beijing, China) with the SyncVR Relax & Distract application (SyncVR, Utrecht, the Netherlands).
  Arms: ICU-VR

SUMMARY:
Rationale: A substantial proportion of the Intensive Care Unit (ICU) survivors develop psychological impairments due to their ICU admission. Several interventions to mitigate these impairments have been explored but lack a proper effect. Intensive Care Unit-specific Virtual Reality has proven to be potentially effective in treating PTSD and depression-related sequelae in ICU-survivors.

Objective: To evaluate the contribution in terms of information provision and patients' perspectives of ICU-VR to prepare lung transplant patients for their future ICU admission

Study design: A monocentre randomized controlled study

Study population: Lung transplant patients who are on the waiting list and understand the Dutch language. Due to the criteria for lung transplantation, these are 18-71 years of age. Participants need to have signed the informed consent formular.

Intervention: The ICU-VR intervention is designed by an interdisciplinary team of intensivists, ICU nurses, a psychiatrist, a psychologist, and a former ICU patient, to expose patients to the ICU environment while offering treatment- and department-related information. During the 12-minute lasting intervention, patients experience different facets of ICU treatment and receive information on the ICU environment, treatment, and workflow. The intervention group will receive this treatment during the appointment with the lung transplantation nurse. The control group will receive the regular hospital preparation care.

Primary endpoints: The primary endpoint will be the difference in information provision of the ICU care of lung transplant patients on the waiting list.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Be on the waiting list for lung transplantation
* Age 18-71 years (maximum age for lung transplantation is 71 years)
* Understand the Dutch language
* Signed informed consent

Exclusion Criteria:

While patients on the waiting list for lung transplantation are intensively monitored and only placed on the waiting list under strict conditions, no additional exclusion criteria above these are identified to exclude specific patients.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percieved quality of information provision | Participants will be followed from inclusion until two weeks after ICU admission, when they complete the last questionnaires.
  The primary endpoint will be the difference in the patients' perceived quality of information provision during preparation of the future planned ICU admission between the intervention and control group, measured after ICU admission. This will be assessed using a subset of the Consumer Quality Index-Relatives ICU (CQI-Relatives ICU), carefully tailored to the needs of this study by members of the RATE-XR steering group and currently being used in another randomized controlled trial investigating the effect of ICU-VR on information provision in relatives of ICU patients. The CQI-Relatives ICU was designed according to a robust method developed by the Healthcare Institute of the Netherlands.

SECONDARY OUTCOMES:
Patients' perspectives and satisfaction with ICU care and the VR intervention | Participants will be followed from inclusion until two weeks after ICU admission, when they complete the last questionnaires.
  Patients' perspectives and satisfaction towards the ICU-VR intervention (only in the intervention group) and perspectives and satisfaction towards the preparation for ICU admission, the delivered ICU care, and the ICU aftercare. This will be measured two weeks after the VR session and two weeks after an ICU discharge using a questionnaire, which was based on the Patient Satisfaction Questionnaire and Family Satisfaction with ICU Care tools. This questionnaire is carefully tailored to the needs of the study, in which we also added some items to evaluate patients' perspectives on the ICU-VR intervention. This questionnaire was previously used in another RCT to evaluate the effect of ICU-VR in post-ICU patients and is currently being used in our HORIZON-IC study (as mentioned in the introduction and rationale)
PTSD | Participants will be followed from inclusion until two weeks after ICU admission, when they complete the last questionnaires.
  The severity of PTSD-related symptoms will be expressed as the sum score of the Impact of Event Scale - Revised (IES-R) and the prevalence of probable PTSD will be expressed as the proportion of patients having an IES-R sum score above 23. The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events. It is a revised version of the older version, the 15-item IES. The IES-R contains seven additional items related to the hyperarousal symptoms of PTSD, which are not included in the original IES. Items are rated on a 5-point scale ranging from 0 ('not at al') to 4 ('extremely'). The IES-R yields a total score (ranging from 0 to 88; higher scores indicate more severe symptoms), and subscale scores can also be calculated for the Intrusion, Avoidance and Hyperarousal subscales. The severity and prevalence of PTSD will be assessed two weeks after an ICU discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands